CLINICAL TRIAL: NCT05244291
Title: The Effect of Therapeutic Touch at Different Times on Colic Symptoms in Infants With Infantile Colic According to Watson's Theory of Human Care: A Randomized Controlled Study
Brief Title: Effect of Therapeutic Touch at Different Times on Infantile Colic According to Watson's Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Karamanoğlu Mehmetbey University, Faculty of Health Science, Pediatric Nursing Department, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 05-2021/27
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Infantile Colic; Therapeutic Touch
Keywords: Therapeutic Touch; infantile colic; infant; Watson's Theory of Human Care; symptom; nursing
MeSH Terms: conditions — Colic | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a single-blind, randomized controlled trial.
Who Masked: Participant
Masking Description: Single blind will be done in the study. Only parents will be blinded. Two weeks follow up will be done in both groups. Since the researcher should implement the intervention, evaluate and manage the process, it will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group 1 (Experimental): Therapeutic Touch will be applied to infants for 3 consecutive days, once a day, 10 minutes at any time during the day. There will be a four-day break. The Therapeutic Touch will be done a total of 3 times in 1 weeks.
  Interventions: Other: Therapeutic Touch
- Intervention Group 2 (Experimental): Therapeutic Touch will be applied to infants for 3 consecutive days, once a day, 10 minutes at any time during the day. There will be a four-day break. The Therapeutic Touch will be done a total of 6 times in 2 weeks.
  Interventions: Other: Therapeutic Touch
- Control Group (No Intervention): The therapeutic touch will not be applied to the control group infants. However, the routine follow-up and behavior of the weekly baby will be evaluated to ensure that parents are blind.

INTERVENTIONS:
Other: Therapeutic Touch — Therapeutic Touch will be applied to infants for 3 consecutive days, once a day, 10 minutes at any time during the day. There will be a four-day break. The Therapeutic Touch will be done a total of 3 times a week or 6 times in 2 weeks.
  Arms: Intervention Group 1; Intervention Group 2

SUMMARY:
Aim: The purpose of the study is to determine the effect of therapeutic touch applied to infants with infantile colic at different times on infant colic scale score, crying and sleep duration, according to Watson's theory of human care. Thus, it is aimed to contribute to the development of an effective care approach in eliminating or reducing the symptoms in infants with infantile colic.

Method: The study will be conducted as a single-blind, randomized controlled trial. The population of the study will be infants who come to the Pediatrics Outpatient Clinic and are diagnosed as infantile colic according to the evaluation of the pediatrician and have no other health problems. The infants will be divided into three groups as intervention (The first group; the group in which therapeutic touch was applied for one week and the second group; the group in which the therapeutic touch was applied for two weeks) and control groups according to stratified block randomization in the computer environment. After the randomization, therapeutic touch will be applied to the intervention group. No method will be applied to the control group.

DETAILED DESCRIPTION:
The research will be carried out with three groups as intervention (The first group; the group in which therapeutic touch was applied for one week and the second group; the group in which the therapeutic touch was applied for two weeks) and control groups. Sample size of the study has been determined by the power analysis, in line with the results obtained from the studies which have been conducted using a similar research method. According to the analysis results, it has been calculated as 32 for each group and 96 in total. Mothers of the infants meeting the study inclusion criteria will be informed both in written and verbally. Written consent will be obtained. The infants will be divided into three groups according to block randomization in the computer environment. The randomization, therapeutic touch will be applied to the intervention group (The first group; the group in which therapeutic touch was applied for one week and the second group; the group in which the therapeutic touch was applied for two weeks). No method will be applied to the control group by the researcher. In obtaining research data, 4 tools will be used: "Mother-infant Information Form", "Infantile Colic Scale", Crying Time Registration Form and Sleep Time Registration Form.

ELIGIBILITY:
Inclusion Criteria:

* Family volunteering to participate in the research
* The infant was born at term
* The infant is between 4 weeks and 8 weeks
* The birth weight is between 2500-4500 g
* The infant has been diagnosed with infantile colic by a physician
* Mothers' ability to read, write and speak Turkish
* New diagnosis of infantile colic

Exclusion Criteria:

* The baby has any chronic disease
* The baby has a congenital anomaly
* The mother has a diagnosed mental and mental problem
* Mother's smoking
* The diagnosis of infants with lactose intolerance by the physician

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Crying Time | In eight weeks.
  Infants' weekly crying times will be recorded (Every day of the week). Weekly crying time will be taken.
Sleeping Time | In eight weeks.
  Infants' weekly sleeping times will be recorded (Every day of the week). Weekly sleeping time will be taken.

SECONDARY OUTCOMES:
Infantile Colic Scale | In eight weeks.
  Ellet et al. (2002) developed a Likert-type scale to determine the factors causing colic and to diagnose colic. Cetinkaya and Başbakkal (2007) tested the validity and reliability of the scale for the Turkish population. The scale consists of 5 sub-dimensions and 19 items.The low total score average from the scale indicates that the colic decreases, and the high average score indicates that the colic increases. Infantile colic scale will be applied to all babies in the study when they complete these weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, Res. Assist. Dr., Principal Investigator — Karamanoğlu Mehmetbey University; Emine Geçkil, Professor, Study Director — Necmettin Erbakan University
Locations (1):
- Karaman Education and Research Hospital, Karaman, Turkey (Türkiye)